CLINICAL TRIAL: NCT00589329
Title: Antibiotics and the Prolongation of Pregnancy in Preterm Labor With an Advanced Cervical Exam
Status: Terminated | Phase: Not Applicable | Type: Interventional
Why Stopped: published data suggest potential harm in other investigations.
Sponsor: MetroHealth Medical Center (Other)
Responsible Party: Principal Investigator, Ted Waters, MFM attending, metroheatlh, MetroHealth Medical Center
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Prevention
Other Study IDs: IRB01-00012
Record Dates: First submitted 2007-12-27; First posted 2008-01-09 (Estimated); Results first posted 2019-09-04 (Actual); Last update posted 2019-09-04 (Actual); Status verified 2019-08

CONDITIONS: Length of Pregnancy Prolongation in Hours
Keywords: Preterm birth; antibiotics; preterm labor; respiratory distress; pergnancy
MeSH Terms: conditions — Premature Birth; Obstetric Labor, Premature; Dyspnea | interventions — Erythromycin; Metronidazole; Anti-Bacterial Agents

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- A (Experimental): roup A will be assigned to receive antibiotics:
  * Erythromycin 250 mg IV q 6 hours x 8 doses, followed erythromycin 250 mg tabs, 1 PO q 8 hours for five days.
  * Metronidazole, 1 gm IV loading dose followed by 500 mg IV q 12 hours x 4 doses, followed by metronidazole 500 mg tabs, 1 PO q 8 hours for five days.
  Interventions: Drug: erythromycin and metronidazole (antibiotics)
- B (Placebo Comparator): Group B will not receive antibiotics for pregnancy prolongation, but will receive a matching masked placebo (IV saline and pill) regimen.
  Interventions: Drug: placebo

INTERVENTIONS:
Drug: erythromycin and metronidazole (antibiotics) — Erythromycin 250 mg IV q 6 hours x 8 doses, followed erythromycin 250 mg tabs, 1 PO q 8 hours for five days.
  Metronidazole, 1 gm IV loading dose followed by 500 mg IV q 12 hours x 4 doses, followed by metronidazole 500 mg tabs, 1 PO q 8 hours for five days
  Arms: A
Drug: placebo — IV and pill placebo
  Arms: B

SUMMARY:
Preterm birth remains a major health concern affecting up to 12% of all live births prior to 37 weeks gestation. As preterm birth can often be associated with infection our proposal is to evaluate in a randomized fashion antibiotics for women with advanced cervical exams.

DETAILED DESCRIPTION:
Preterm birth, its causes, prevention, complications and ramifications persist as an important focus of obstetrical research. In the United States 11.8% of all live births occur prior to 37 weeks gestation. As many as 45% of these deliveries will have been proceeded by preterm labor with intact membranes.(2) Both preterm labor and preterm premature rupture of membranes have both been associated with evidence intrauterine infection. While antibiotic treatment in conservative management of preterm PROM remote from term has been shown to significantly prolong pregnancy and reduce infant morbidity, (16) data regarding the effectiveness of antibiotics for pregnancy prolongation in preterm labor are inconsistent. (3-15) Currently, narrow spectrum antibiotics (penicillin or clindamycin) are given prior to delivery to reduce the risk of neonatal Group B Beta Streptococcus (GBS) sepsis, however broad spectrum antibiotic treatment of women with preterm labor for pregnancy prolongation is not recommended.

Review of the literature regarding antibiotic treatment for pregnancy prolongation in preterm labor reveals that most studies utilized single agent therapy, and no study has evaluated the use of antibiotics for pregnancy prolongation in women with an advanced cervical exam (>4cm). While a number of studies have shown significant pregnancy prolongation in unselected populations,(5,12,13) only one study of 12 reviewed was able to show a neonatal benefit to adjunctive antibiotic use.(12,20) Norman, et al was able to show a reduction in the incidence of necrotising enterocolitis with the use of antibiotics. Given the number of studies in this area, and the lack of supporting evidence, this likely represents an alpha error. Another study by Svare et al was able to show a significant decrease in NICU admissions for women treated with antibiotics in the setting of preterm labor, however no change was reported in neonatal morbidities.

Our proposed study is designed to evaluate patients at particular risk for preterm delivery; those with advanced cervical exam. In this randomized prospective controlled study, we intend to examine the influence of adjunctive antibiotic use in preterm labor complicated by a cervical exam of 4 cm or greater. We plan to compare a study group receiving broad-spectrum antibiotics with a control group that will not receive antibiotics for pregnancy prolongation. Both groups will receive antibiotics for GBS prophylaxis as indicated. We hope to see a delay in delivery in the study group as a primary outcome. Secondary outcomes will include the use of steroids, neonatal complications including sepsis, intraventricular hemorrhage, periventricular leukomalacea, mechanical ventilation and respiratory distress syndrome, retinopathy of prematurity and necrotizing enterocolitis, and neonatal ICU stay.

ELIGIBILITY:
Inclusion Criteria:

1. All patients admitted with the diagnosis of preterm labor between 24 0/7 and 33 6/7 weeks gestation. Preterm labor will be defined by regular contractions and/or cervical change from last documented exam.
2. Cervical exam 4 cm or greater
3. Intact membranes

Exclusion Criteria:

1. Multiple gestation (>2)
2. Clinical evidence of chorioamnionitis, such as maternal fever, uterine tenderness, fetal tachycardia
3. Lethal fetal anomaly
4. Persistent vaginal bleeding, abruption, or placenta previa
5. Rupture of membranes
6. Maternal illness or fetal indication requiring delivery
7. Inability to give informed consent
8. Serious allergy to study medications. GI discomfort will not be considered a drug allergy

Ages: 18 Years to 40 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 20 (Actual)
Dates: Start 2007-12; Primary Completion 2012-10 (Actual); Study Completion 2012-10 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Brian Mercer, M.D., Principal Investigator — MetroHealth Medical Center MFM Director; Thaddeus Waters, M.D., Principal Investigator — MetroHealth Medical Center
Locations (1):
- MetroHealth Medical Center, Cleveland, Ohio, United States

RESULTS

PARTICIPANT FLOW:
Groups:
- Group A: Group A will be assigned to receive antibiotics:
  * Erythromycin 250 mg IV q 6 hours x 8 doses, followed erythromycin 250 mg tabs, 1 PO q 8 hours for five days.
  * Metronidazole, 1 gm IV loading dose followed by 500 mg IV q 12 hours x 4 doses, followed by metronidazole 500 mg tabs, 1 PO q 8 hours for five days.
  erythromycin and metronidazole (antibiotics): Erythromycin 250 mg IV q 6 hours x 8 doses, followed erythromycin 250 mg tabs, 1 PO q 8 hours for five days.
  Metronidazole, 1 gm IV loading dose followed by 500 mg IV q 12 hours x 4 doses, followed by metronidazole 500 mg tabs, 1 PO q 8 hours for five days
- Group B: Group B will not receive antibiotics for pregnancy prolongation, but will receive a matching masked placebo (IV saline and pill) regimen.
  placebo: IV and pill placebo
Period: Overall Study
Arm/Group | Group A | Group B
Started | 10 | 10
Completed | 10 | 10
Not Completed | 0 | 0

BASELINE CHARACTERISTICS:
Groups:
- Group A: Antibiotic group
- Group B: Non antibiotic group
- Total: Total of all reporting groups
Arm/Group | Group A | Group B | Total
Number analyzed (Participants) | 10 | 10 | 20
Age, Customized [Count of Participants; unit: Participants] | 10 | 10 | 20
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 10 | 10 | 20
  Male | 0 | 0 | 0
Region of Enrollment [Number; unit: participants]
  United States | 10 | 10 | 20

OUTCOME MEASURES:

1. Primary Outcome: Length of Pregnancy Prolongation
Description: The length of time (in hours) from initiation of therapy to delivery will establish the latency
Time Frame: Measured from randomization to delivery in hours
Measure: Mean (Full Range); unit: hours
Arm/Group | Group A | Group B
Number analyzed (Participants) | 10 | 10
hours | 4 [0 to 36] | 4 [1 to 38]

2. Secondary Outcome: Respiratory Distress
Description: Respiratory distress will be defined by the clinical record documentation of the neonatal team.
Time Frame: newborn nursery
Measure: Count of Participants; unit: Participants
Groups:
- Group A: roup A will be assigned to receive antibiotics:
  * Erythromycin 250 mg IV q 6 hours x 8 doses, followed erythromycin 250 mg tabs, 1 PO q 8 hours for five days.
  * Metronidazole, 1 gm IV loading dose followed by 500 mg IV q 12 hours x 4 doses, followed by metronidazole 500 mg tabs, 1 PO q 8 hours for five days.
  erythromycin and metronidazole (antibiotics): Erythromycin 250 mg IV q 6 hours x 8 doses, followed erythromycin 250 mg tabs, 1 PO q 8 hours for five days.
  Metronidazole, 1 gm IV loading dose followed by 500 mg IV q 12 hours x 4 doses, followed by metronidazole 500 mg tabs, 1 PO q 8 hours for five days
Arm/Group | Group A | Group B
Number analyzed (Participants) | 10 | 10
Participants | 2 | 1

ADVERSE EVENTS:
Arm/Group | Group A | Group B
Serious Adverse Events (participants affected / at risk) | 0/10 | 0/10
Other Adverse Events (participants affected / at risk) | 0/10 | 0/10

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes